CLINICAL TRIAL: NCT01479751
Title: Comparison of Mg, Ketamine, Large Dose Rocuronium, and Priming on Intubating Condition in Rapid Sequence Intubation
Brief Title: Comparison of Methods to Facilitate Rapid Sequence Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Kim Mihyun, clinical professor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: facilitating RSI
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2012-08-27 (Estimated); Status verified 2012-08

CONDITIONS: Intubating Condition
Keywords: Rocuronium; magnesium; priming; ketamine; intubation
MeSH Terms: interventions — Magnesium Sulfate; Ketamine; Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- ketamine (Experimental): Patients receive ketamine 0.5 mg/kg 2 min before Roc injection.
  Interventions: Drug: Ketamine
- priming (Experimental): Patients receive Roc 0.06 mg/ kg as a priming dose 3 min before injection of Roc 0.54 mg/kg.
  Interventions: Drug: rocuronium
- Roc 0.9 (No Intervention): Patients receive Roc 0.9 mg/kg as an induction dose.
- Control (No Intervention): Patients receive Roc 0.6 mg/kg without any pretreatments of Mg, ketamine, or priming.
- Mg (Experimental): Patients receive magnesium sulfate (MgSO4) 50 mg/kg over 10 min before Roc injection.
  Interventions: Drug: Magnesium Sulfate

INTERVENTIONS:
Drug: Magnesium Sulfate — Patients receive MgSO4 50 mg/kg for 10 min before injection of Roc 0.6 mg/kg.
  Arms: Mg
Drug: Ketamine — patients receive ketamine 0.5 mg/kg 2 min before Roc injection.
  Arms: ketamine
Drug: rocuronium — Patients receive Roc 0.06 mg/ kg as a priming dose 3 min before injection of Roc 0.54 mg/kg.
  Arms: priming

SUMMARY:
In this study, methods which are known for facilitating rapid sequence intubation or accelerating rocuronium (Roc)onset are compared including magnesium (Mg), ketamine pretreatment, large dose rocuronium and priming.

DETAILED DESCRIPTION:
Patients are pretreated with Mg, ketamine, or priming dose Roc. Two groups do not receive pretreatment, but are given Roc 0.6 mg/kg or 0.9 mg/kg.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 65 years,
* ASA 1 - 2,
* patients scheduled for elective surgery under general anesthesia,
* BMI 18.5-24.9 kg/m2
* Mallampati class I-II

Exclusion Criteria:

* neuromuscular disorder,
* cardiac/hepatic/renal insufficiency,
* pregnant.
* anticipated difficult airway
* medications that influence neuromuscular transmission

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Intubation score | participants will be followed at the time point of intubation, an expected average of 70 sec from the start of rocuronium injection.
  Patients are tracheally intubated, and intubation scores(poor, good,excellent)are rated.

SECONDARY OUTCOMES:
Roc duration | participants will be followed when TOF count reaches two, an expected average of 40 min.
  Time from the start of rocuronium injection until reappearance of two muscle twitches in TOF stimulations is measured, using ToF-Watch sx.
Roc onset | participants will be followed when TOFcount =0 within an expected average of 4 min from the start of rocuronium injection.
  Time from the start of rocuronium injection until TOF count=0 using TOF-Watch sx.
Hemodynamic variables | participants will be followed at baseline, before and for 5 min after the intubation, an expected average of 8 min after the start of anesthetic induction.
  Mean arterial pressure (MAP)and heart rate (HR) are measured at baseline, before intubation, and 1, 2, 3, 4, 5 min after intubation.
TOF% at intubation | participants will be followed at the time point of intubation, an expected average of 70 sec from the start of rocuronium injection.
  neumeric value expressed as %, displayed on the monitor of TOF watch-Sx in TOF stimulation (ex. 5% on the display means 95% suppression of T1)

CONTACTS AND LOCATIONS:
Overall Officials: Mihyun Kim, doctor, Principal Investigator — Seoul National University Bundang Hospital
Locations (1):
- Seoul National University Bundang hopital, Seongnam-si, Gyeonggi-do, South Korea